CLINICAL TRIAL: NCT04044976
Title: Treatment With Caffeine of Very Preterm Infant in the Delivery Room: the CAFROOM Feasibility Study
Brief Title: Caffeine Treatment in in the Delivery Room
Acronym: CAFROOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Carlo Dani, Full Professor of Pediatrics, University of Florence
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 02/2019
Record Dates: First submitted 2019-07-30; First posted 2019-08-05 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Distress Syndrome
Keywords: Caffeine; delivery room; preterm infant
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — caffeine citrate; Caffeine

STUDY DESIGN:
Intervention Model Description: A cohort of preterm infants will be given caffeine in the delivery room
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated infants (Experimental): Infants who will receive caffeine in the delivery room.
  Interventions: Drug: Caffeine Citrate

INTERVENTIONS:
Drug: Caffeine Citrate — Infants will receive 20 mg/kg of caffeine citrate intravenously, via the umbilical vein, or enterally, through an orogastric tube, within 10 min of birth.
  Other Names: Caffeine

SUMMARY:
Background. In recent years, particular attention has been paid to all interventions that could help reduce the need for mechanical ventilation MV and, therefore, the risk of BPD. However, early application of non-invasive respiratory supports and early treatment with surfactant fail in 45-50% of cases. Failure frequently depends on the onset of apnea episodes and, therefore, it has been proposed to treat very preterm infants with caffeine already in the delivery room in the first min of life.

Hypothesis and objectives of the study. Our aim is to verify the hypothesis that it is possible to administer caffeine in the delivery room intravenously and enterally via an orogastric tube.

Study design. Infants 25-29 weeks of gestational age will be enrolled and will be randomized to receive 20 mg/kg of caffeine citrate intravenously, via the umbilical vein, or enterally, through an orogastric tube, within 10 min of birth. The dosage of plasma caffeine concentration will be performed 60+15 min after administration to measure its peak and 60+15 min before the next dose (5 mg/kg/day i.v.).

Endpoints. The primary endpoint will be the evaluation of the success rate of intravenous or enteral administration of caffeine in the delivery room. Secondary endpoints will be the evaluation of: number of infants in whom caffeine will be successfully administered by intravenous versus enteral route; number of infants where caffeine will be successfully administered that reached the therapeutic plasmatic range the first dose, confirming the success of the administration; comparison of caffeine blood level obtained with intravenous and enteral administration; frequency of successes in obtaining the therapeutic range after the second dose; frequency of MV within the first 72 hours of life in studied infants.

Statistical analysis. In the absence of previous studies to use as a reference and this study being a feasibility study, it was decided arbitrarily to study 20 infants treated in the delivery room with caffeine administered intravenously and 20 infants treated in the delivery room with caffeine administered enterally. The clinical characteristics of the two groups will be described by calculating the mean value and the standard deviation or the rate and percentage. The primary endpoint will be evaluated by calculating the percentage of cases in which caffeine will be successfully administered. The comparison between the number of infants in which caffeine will be successfully administered intravenously versus the enteral route and the comparison between the caffeine plasma level obtained with intravenous and enteral administration will be performed using the Student "t" test for continuous parametric variables, the Wilcoxon rank sum test for non-parametric continuous variables and the χ2 test for categorical variables. A p <0.05 will be considered as statistically significant.

DETAILED DESCRIPTION:
INTRODUCTION Background Mechanical ventilation (MV) is one of the most important risk factors for the development of bronchopulmonary dysplasia (BPD) in the preterm infant, due to the early pulmonary inflammation from volume- and baro-trauma and the secondary 1. Despite this, around 80% of infants born with gestational age <27 weeks must be treated with MV 2 for a respiratory distress syndrome (RDS), and in about 65% of cases it starts already in the delivery room in the first min of life 3.

Therefore, in recent years particular attention has been paid to all interventions that could help reduce the need of MV, thus reducing the risk of BPD. Among these interventions, the early application of non-invasive continuous positive airway pressure (CPAP), the use of sustained lung inflation (SLI), and early treatment with surfactant with INSurE (Intubation- Surfactant-Extubation) or LISA (less invasive surfactant administration) 1,4. These interventions have the common objective of promoting lung recruitment by promoting the development and maintenance of alveolar residual functional capacity (CFR), improving pulmonary compliance, reducing work of breathing and favoring gas exchange 1,4. Unfortunately, these treatments are not always effective and recent studies have shown that CPAP in combination or not with surfactant administration fails to prevent MV in about 45-50% of treated infants 3; similarly the SLI strategy in association with non-invasive CPAP and with the possible administration of surfactant fails to prevent MV in approximately 60% of treated infants 5. In fact, in many cases the failure of MV prevention does not depend on severity of RDS, which also remains a very important factor, but especially in mild-moderate forms of RDS is due to the onset of relapsing episodes of apnea. Therefore, it has been proposed to treat very preterm infants with caffeine in the delivery room already in the first min of life. This drug is very effective in the preterm infant in whom it has been shown to decrease the frequency of apnea, the risk of BPD, the duration of non-invasive respiratory supports, and the risk of re-intubation 6, also in infants without previous crisis of apnea 7.In fact, caffeine stimulates spontaneous respiratory activity, improves lung compliance and minute volume, reduces airway resistance, and increases diaphragm contractility, together with a good safety profile and without significant side effects at current doses 6. In a recent pilot study, Katheria et al. randomized 21 infants with gestational age <29 weeks to receive 20 mg/kg of caffeine citrate within 2 h of life or at 12 hours of life obtaining in treated infants a decrease, although not statistically significant, of the need of VM (27 vs. 70%) in association with an overall hemodynamic improvement 8. Subsequently, Dekker et al. randomized 23 infants of 24-29 gestational weeks to receive 10 mg/kg of caffeine in the delivery room or immediately after arrival in neonatal intensive care unit (4.4 vs. 48 min of life) demonstrating that early treatment is associated with a significant increase in tidal volume and a lower need for oxygen-therapy 9. Although the results were promising, neither study measured the plasma concentration of caffeine or had sufficient statistical power to assess whether caffeine administered in the delivery room is effective in reducing the risk of mechanical ventilation.

Study hypothesis The present feasibility study aims to evaluate the possibility of administering caffeine in the delivery room intravenously and enterally through an orogastric tube during the postnatal stabilization of the preterm infant. It is preliminary to the planning of a subsequent randomized controlled trial of adequate size, which will aim to assess whether caffeine administered so early can actually reduce the risk of MV in preterm infants.

Objectives of the study Primary objectives of the study. The primary objective will be the evaluation of the feasibility of the administration of intravenous or enteral caffeine in the very preterm infant in the delivery room during assistance for cardiorespiratory stabilization of the infant.

Secondary objectives of the study. The secondary objectives will be to compare the feasibility of administering caffeine intravenously vs. enteral and evaluation of the need for MV in treated infants.

MATERIALS AND METHODS Patients. The study will be conducted in 2 Third Level Neonatal Intensive Care Units after approval by local ethics committees.

Inclusion criteria. Once the written informed consent of the parents or legal guardians has been obtained, inborn infants of 25+0-29+6 weeks of gestational age at high risk of developing "respiratory distress syndrome" (RDS), who do not require MV in the delivery room, will be enrolled in the study.

Exclusion criteria. Exclusion criteria will be: maternal consumption of caffeine before giving birth (> 2 cups of coffee in the 6 hours before birth), major congenital malformations, chromosomal syndromes, fetal hydrops, and inherited metabolic disorders.

Design of the study. Infants will be electronically randomized to receive 20 mg/kg (1 mL=20 mg) of caffeine citrate (Peyona®, Chiesi Farmaceutici Spa, Parma, Italy) intravenously, via the umbilical vein, or enterally, through an orogastric tube, within 10 min of birth.

Intravenous administration may take place via an umbilical venous catheter or a "butterfly" needle inserted into the umbilical vein. The bolus of caffeine will be followed by the administration of a 2 mL "flush" of saline both in the case of administration by venous and enteral route. Successes and failures of the administration with the two different methods will be recorded.

The level of plasma caffeine concentration will be measured 60+15 min after the administration to evaluate its peak and 60+15 min before the administration of the second dose (5 mg/kg/day i.v.) which will be given after admission in neonatal intensive care unit 10. The plasma level will be measured using the "dried blood spots" method with spectrometry and "tandem-mass" liquid chromatography 11 in the Laboratory of Clinical Chemistry and Pharmacology of the A. Meyer Pediatric Hospital of Florence. Blood samples will be collected with heel punctures commonly performed for monitoring these patients and stored at -80°C until to analysis.

If necessary, resuscitation in the delivery room will be performed following the guidelines of the AAP/ AAH 12. After admission in neonatal intensive care, infants who have not required VM in the delivery room will be assisted with the following non-invasive respiratory supports: nasal continuous positive airway pressure (NCPAP), "bi-level" NCPAP (BiPAP), nasal intermittent mandatory ventilation (N-IMV) using a CDP/ PEEP of 5-8 cmH2O. Surfactant (Curosurf ®, Chiesi, Parma, Italy) will be given (200 mg/kg) according to the INSURE (Intubation-SURfactant-Extubation) or LISA (Less-Invasive-Surfactant-Administration) technique in infants requiring FiO2 >0.30 to maintain a SpO2 90-95% and in all infants who will need MV.

MV will be started in the case of pCO2 >65 mmHg and pH <7.20, or pO2 <50 mm Hg with FiO2 >0.50 after surfactant administration or in case of apnea (> 4 episodes in 1 hour or> 2 episodes in 1 hour requiring manual ventilation), and will be conducted with the aim of maintaining a pCO2 of 55-65 mmHg and a SpO2 of 90-95% 9, using synchronized VM (patient triggered ventilation: PTV), or the volume controlled VM, or high frequency ventilation (HFV).

Collected data. For each infant will be recorded: gestational age; birth weight; birth weight <10th percentile; gender; type of delivery; Apgar score at 5 min; main disorders of pregnancy (pre-eclampsia, premature rupture of membranes, clinical chorioamniositis, placental abruption); RDS, whose diagnosis will be based on the occurrence of oxygen-dependence, tachypnea, dyspnea, exclusion of other causes of respiratory failure, and the presence of a typical radiological pattern; treatment with surfactant and nitric oxide; need, type and duration of respiratory assistance (oxygen therapy, NCPAP, BiPAP, N-IMV, PTV, HFV); prenatal and postnatal steroid treatment. In addition, common complications of prematurity will be recorded: patency of the ductus arteriosus (PDA) requiring drug therapy, bronchopulmonary dysplasia (BPD), intraventricular hemorrhage (ICH) of 3-4 grade 13, periventricular leukomalacia (LPV) 14, retinopathy of prematurity (ROP) of grade >3 15, necrotizing enterocolitis (NEC) <2 grade 16, and sepsis. In addition, mortality and the duration of hospitalization will be reported.

Permitted concomitant pharmacological treatments. The enrolled patients can be treated with the following drugs: surfactant, caffeine, doxapram, ibuprofen, paracetamol, indomethacin, dopamine, dobutamine, milrinone, adrenaline, diuretics, antibiotics, glucocorticoids, immunoglobulins, antiepileptics, nitric oxide, analgesics, sedatives.

List of participating centers. Patients will be enrolled at the neonatal intensive care units of Careggi University Hospital of Florence and of IRCCS Foundation - Ospedale Maggiore Policlinico Mangiagalli and Regina Elena of Milan.

ENDPOINTS Primary endpoint. The primary endpoint will be the evaluation of the number of infants in whom the administration of caffeine intravenously or enterally will occur successfully in the delivery room delivery within 10 min of life.

Secondary endpoints. Secondary endpoints will be the evaluation of: number of infants in whom caffeine will be successfully administered by intravenous versus enteral route; number of infants where caffeine will be successfully administered that reached the therapeutic plasmatic range the first dose, confirming the success of the administration; comparison of caffeine blood level obtained with intravenous and enteral administration; frequency of successes in reaching the therapeutic range after the second dose; frequency of VM within the first 72 hours of life in studied infants.

STATISTICAL ANALYSIS Sample size. In the absence of previous studies to use as a reference and this study being a feasibility study, it was decided arbitrarily to study 20 infants treated in the delivery room with caffeine administered intravenously and 20 infants treated in the delivery room with caffeine administered enterally.

Description and analysis of data. The clinical characteristics of the two groups will be described by calculating the mean value and the standard deviation or the rate and percentage.

The primary endpoint will be evaluated by calculating the percentage of cases in which caffeine will be successfully administered. Similarly, the secondary endpoints, represented by the number of cases in which the therapeutic plasmatic range will be reached after the first and the second dose of caffeine and the frequency of VM within the first 72 hours of life, will be evaluated. The comparison between the number of infants in which caffeine will be successfully administered intravenously versus the enteral route and the comparison between the caffeine plasma level obtained with intravenous and enteral administration will be performed using the Student "t" test for continuous parametric variables, the Wilcoxon rank sum test for non-parametric continuous variables and the χ2 test for categorical variables. A p <0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infants
* Infants with 25+0-29+6 weeks of gestational age
* Infants who do not require MV in the delivery room

Exclusion Criteria:

* Maternal consumption of caffeine before giving birth (> 2 cups of coffee in the 6 hours before birth)
* Major congenital malformations
* Chromosomal syndromes
* Fetal hydrops
* Inherited metabolic disorders

Ages: 1 Minute to 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Successful rate | 10 minutes after birth
  Evaluation of the number of infants in which the administration of intravenous or enteral caffeine in the delivery room will occur successfully

SECONDARY OUTCOMES:
Comparison of intravenous versus enteral route | 10 minutes after birth
  Evaluation of number of infants in whom caffeine will be successfully administered by intravenous versus enteral route
Caffeine administration and its therapeutic range | 90 minutes after birth
  Number of infants in whom caffeine will be successfully administered that reached the therapeutic plasmatic range after the first dose
Intravenous vs enteral caffeine administration and therapeutic range | 90 minutes after birth
  Comparison of caffeine blood level obtained with intravenous and enteral administration
Need of mechanical ventilation | 72 hours of life
  Frequency of VM in studied infants

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Neonatology, Careggi University Hospital, Florence, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected in electronic sheet. These data will be available on request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available at the end of the study.
Access Criteria: Access will be allowed on request.

REFERENCES:
- [Derived] Dani C, Cecchi A, Ciarcia M, Miselli F, Luzzati M, Remaschi G, Bona MD, la Marca G, Boni L. Enteral and Parenteral Treatment with Caffeine for Preterm Infants in the Delivery Room: A Randomised Trial. Paediatr Drugs. 2023 Jan;25(1):79-86. doi: 10.1007/s40272-022-00541-y. Epub 2022 Oct 27. PMID 36301511
- [Derived] Dani C, Cecchi A, Remaschi G, Mercadante D, la Marca G, Boni L, Mosca F. Study protocol: treatment with caffeine of the very preterm infant in the delivery room: a feasibility study. BMJ Open. 2020 Dec 4;10(12):e040105. doi: 10.1136/bmjopen-2020-040105. PMID 33277284